CLINICAL TRIAL: NCT01635959
Title: Prevalence of Gastroesophageal Reflux Disease (GERD) in Patients With Upper Gastrointestinal Tract Symptoms in Egypt
Acronym: GERD Q NIS
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-GEG-XXX-2012/1
Record Dates: First submitted 2012-07-03; First posted 2012-07-10 (Estimated); Last update posted 2014-10-03 (Estimated); Status verified 2014-10

CONDITIONS: Patients With Upper Gastro-intestinal Symptoms
Keywords: upper gastro-intestinal symptoms, GERD
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with Gastrointestinal Trackt Symptoms

SUMMARY:
The purpose of this study is to calculate the prevalence of gastroesophageal reflux disease (GERD) by mean of GERD-Q questionnaire in patients with upper gastrointestinal tract symptoms in Egypt.

DETAILED DESCRIPTION:
Prevalence of Gastroesophageal reflux disease (GERD) in patients with upper gastrointestinal tract symptoms in Egypt

ELIGIBILITY:
Inclusion Criteria:

* 18 years and above
* Attending the medical office and reporting symptoms suggestive of upper gastrointestinal tract symptoms such as heartburn/regurgitation, abdominal pain, bloating, belching and nausea/vomiting.

Exclusion Criteria:

* Participating on a clinical trial during the last 3 months.
* Patients not able to read and/or understand the GERD-Q questionnaire.
* Patients already included in the study in other participating site.
* Patients taking PPIs or H2blockers in the l

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community patients
Sampling Method: Non-Probability Sample
Enrollment: 3170 (Actual)
Dates: Start 2012-07; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Percentage of patients scoring ≥ 8 in GERD-Q | baseline
  Percentage of patients scoring ≥ 8 in GERD-Q will be considered as suffering from GERD.
  The GERD-Q is a potentially useful tool for family practitioners and other health care professionals in diagnosing and managing GERD without initial specialist referral or endoscopy.
  The Egyptian-validated version of the GERD-Q will be used for the study purposes.

SECONDARY OUTCOMES:
Socio-demographic characteristics of patients diagnosed with gastroesophageal reflux disease (GERD) | baseline
  Descriptive analysis of socio-demographic characteristics of patients diagnosed with gastroesophageal reflux disease (GERD) in Egypt.
Treatment patterns in patients diagnosed with gastroesophageal reflux disease (GERD) | baseline
  Descriptive analysis of treatment patterns in patients diagnosed with gastroesophageal reflux disease (GERD) in Egypt.

CONTACTS AND LOCATIONS:
Overall Officials: Dina A Ahmed, MD, Study Director
Locations (21):
- Egypt (21):
  - Research Site, Al Mansurah
  - Research Site, Al Menia
  - Research Site, Alex
  - Research Site, Asuit
  - Research Site, Aswān
  - Research Site, Banhā
  - Research Site, Cairo
  - Research Site, Domiaat
  - Research Site, Hurghada
  - Research Site, Ismailia
  - Research Site, Kafr ash Shaykh
  - Research Site, Kalubia
  - Research Site, Luxor
  - Research Site, Mahala
  - Research Site, Menofia
  - Research Site, Port-Saeed
  - Research Site, Qina
  - Research Site, Sharkiah
  - Research Site, Sohag
  - Research Site, Suiz
  - Research Site, Tanta